CLINICAL TRIAL: NCT05561140
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy of Voxelotor for the Treatment of Leg Ulcers in Patients With Sickle Cell Disease
Brief Title: Resolution of Sickle Cell Leg Ulcers With Voxelotor
Acronym: RESOLVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Emerging clinical data evaluated by Pfizer and shared with regulatory authorities indicates that the risk profile of voxelotor in people with SCD exceeds the benefits observed in previously generated global research and requires further assessment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GBT440-042; C5341026 (Other: Alias Study Number)
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease; Leg Ulcers
Keywords: Sickle Cell Disease, SCD
MeSH Terms: conditions — Anemia, Sickle Cell; Leg Ulcer | interventions — voxelotor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Voxeletor + SOC (Standard of Care) (Experimental)
  Interventions: Drug: Voxelotor Oral Tablet
- Placebo + SOC (Standard of Care) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Voxelotor Oral Tablet — Synthetic small molecule supplied as 500 mg tablets, administered Orally
  Arms: Voxeletor + SOC (Standard of Care)
Other: Placebo — Placebo
  Arms: Placebo + SOC (Standard of Care)

SUMMARY:
This study is a Phase 3, multicenter, randomized, placebo-controlled study to evaluate the efficacy of voxelotor and standard of care for the treatment of leg ulcers in participants with sickle cell disease. The study is divided into a 5 study periods: Screening, Run-in, Randomized Treatment, Open-label Treatment, and Follow-up/End of Study (EOS).

The study will be conducted in approximately 80 eligible participants at approximately 20 global clinical trial sites.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with documented diagnosis of SCD (HbSS, HbS/β0 thalassemia)
2. Age 12 years and older
3. At least 1 cutaneous ulcer(s) on the lower extremity (leg, ankle, or dorsum of foot) that meets the following criteria:

   * Duration: ≥ 2 weeks and < 6 months at Screening, and
   * Size: > 2 cm2 prior to randomization
4. Written informed consent (≥ 18 years) or parental/guardian consent and participant assent (≥ 12-17 years) per IEC policy and requirements, consistent with ICH guidelines

Exclusion Criteria:

1. Target ulcer(s) healed by ≥ 25% during the standard of care run-in period prior to randomization
2. Active infection/purulence at ulcer site, or exposed tendon or bone at the ulcer site, based on Investigator's clinical judgment
3. Current osteomyelitis at or near the ulcer site
4. Known vascular abnormalities that would preclude healing in the opinion of the Investigator (eg, pre-existing severe arterial insufficiency in the affected limb)
5. Serum albumin < 2.0 g/dL
6. RBC transfusion within 60 days of initiation of study drug
7. Receiving regularly scheduled RBC transfusion therapy (also termed chronic, prophylactic, or preventive transfusion) during the study
8. Planned elective surgery within the next 6 months
9. Anemia due to bone marrow failure (eg, myelodysplasia)
10. Absolute reticulocyte count < 100 × 109/L
11. Screening alanine aminotransferase (ALT) > 4 × upper limit of normal (ULN)
12. Severe renal dysfunction (estimated glomerular filtration rate [eGFR] < 30 mL/min/1.73 m2 by Schwartz formula) or is on chronic dialysis
13. Clinically significant bacterial, fungal, parasitic, or viral infection that requires therapy

Other protocol-defined Eligibility Criteria that apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- Brazil (9):
  - Complexo Hospitalar Universitário Professor Edgard Santos- Universidade Federal Da Bahia, Salvador, Estado de Bahia
  - Universidade Federal Da Bahia Hospital Universitário Professor Edgard Santos, Salvador, Estado de Bahia
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Hospital das Clinicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Multihemo Servicos Medicos S/A, Recife, Pernambuco
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, Cerqueira Cesar - Sao Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Esho Empresa De Servicos Hospitalares S.A/ Hospital Samaritano Higienopolis, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Kenya (6):
  - KEMRI Centre for Clinical Research Butere County Hospital, Butere, Kakamega County
  - KEMRI Kondele Children's Hospital within Jaramogi Oginga Odinga Teaching and Referral Hospital., Kisumu
  - Gertrude's Children's Hospital, Nairobi
  - KEMRI-Centre for Respiratory Diseases Research-Nairobi, Nairobi
  - Strathmore University Medical Centre, Nairobi
  - KEMRI-CRDR, KEMRI Clinical Research Annex, Siaya
- Nigeria (7):
  - SYNLAB, Gwagwalada, Abuja
  - University of Calabar Teaching Hospital, Calabar, Cross River State
  - SYNLAB, Abuja, Federal Capital Territory
  - University of Abuja Teaching Hospital, Gwagwalada, Federal Capital Territory
  - Barau Dikko Teaching Hospital/Kaduna State University, Kaduna
  - Aminu kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lagos

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 88 participants with sickle cell disease (SCD) were enrolled, randomized and treated with study drug for leg ulcers.
Pre-assignment Details: Eligible participants were randomized to receive study drug for 12 weeks in DB randomized period.Following this,eligible participants received voxelotor (delayed) for minimum 12 weeks in OL period. Participants were followed up for 4 weeks after last dose of study drug. All participants received the SOC per investigator/protocol for SCD leg ulcers.
Groups:
- Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC: Participants were randomized to receive voxelotor 1500 milligram (mg) (3 tablets*500 mg) orally once daily (OD) and SOC for 12 weeks in double blinded randomized treatment period. Eligible participants then in open label treatment period, continued to receive voxelotor 1500 mg (3 tablets*500 mg) orally OD and SOC for minimum of 12 weeks.
- Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC: Participants were randomized to receive placebo matched to voxelotor, orally OD and SOC for 12 weeks in double blinded randomized treatment period. Eligible participants then in open label treatment period, received voxelotor 1500 mg (3 tablets*500 mg) orally OD and SOC for minimum of 12 weeks.
Period: Randomized Treatment Period
Arm/Group | Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC
Started | 45 | 43
Completed | 43 | 43
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Open Label Treatment Period
Arm/Group | Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC
Started | 43 | 43
Completed | 5 | 6
Not Completed | 38 | 37
Not completed — Adverse Event | 6 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Study terminated by sponsor | 29 | 30
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC: Participants were randomized to receive voxelotor 1500 mg (3 tablets*500 mg) orally, OD and SOC for 12 weeks in double blinded randomized treatment period. Eligible participants then in open label treatment period, continued to receive voxelotor 1500 mg (3 tablets*500 mg) orally OD and SOC for minimum of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.2 (7.61) | 25.1 (8.53) | 24.64 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 24 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 34 | 28 | 62
  Unknown or Not Reported | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 42 | 87
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Resolution of the Target Ulcers by Week 12 in Randomized Treatment Period
Description: An ulcer qualified as a target ulcer, if met the following criteria: a) duration of ulcer was greater than equal to (>=) 2 weeks and less than (<) 6 months at screening; b) healed by <25 percent (%) during the SOC run-in phase prior to randomization; c) size was greater than (>2) square centimeters (cm^2) at any visit, prior to randomization. Resolution of the target ulcer was defined as skin re-epithelialization confirmed at 2 consecutive study visits, 2 weeks apart during the 12-week randomized treatment period. For participants with more than one target ulcer, all target ulcers must be confirmed resolved in order for the participant to be a responder.
Time Frame: Through Week 12 of randomized treatment period
Population: Intention to treat (ITT) population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC
Number analyzed (Participants) | 45 | 43
Percentage of participants | 6.7 [1.4 to 18.3] | 7.0 [1.5 to 19.1]
Statistical Analysis 1: Comparison: Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC vs Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Difference in percentage = -0.3, 95% CI 2-sided [-10.9 to 10.2]

2. Secondary Outcome: Time to Resolution of Target Ulcers up to Week 12 in Randomized Treatment Period
Description: An ulcer qualified as a target ulcer, if met the following criteria: a) duration of ulcer was >=2 weeks and <6 months at screening; b) healed by <25% during the SOC run-in phase prior to randomization; c) size was >2 cm^2 at any visit, prior to randomization. Resolution of the target ulcer was defined as skin re-epithelialization confirmed at 2 consecutive study visits, 2 weeks apart during the 12-week randomized treatment period. Time to resolution of target ulcers was defined as the first time of the observed ulcer was resolved. For participants with more than one target ulcer, time to resolution of target ulcers was defined as time to the last target ulcer confirmed resolved. For participants who did not have the last target ulcer confirmed resolved by Week 12 or who were discontinued from study, the time to resolution was censored. Median time to event was evaluated using Kaplan-Meier method.
Time Frame: From Day 1 to censoring date before Week 12 or maximum up to Week 12 of randomized treatment period, whichever occurred first
Population: ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC
Number analyzed (Participants) | 45 | 43
Days | NA [NA to NA] — Median and 95% confidence interval (CI) was not estimated due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI was not estimated due to insufficient number of participants with events.

3. Secondary Outcome: Change From Baseline in Total Surface Area of Target Ulcers at Week 12 in Randomized Treatment Period
Description: An ulcer qualified as a target ulcer, if met the following criteria: a) duration of ulcer was >=2 weeks and <6 months at screening; b) healed by <25% during the SOC run-in phase prior to randomization; c) size was >2 cm^2 at any visit, prior to randomization.
Time Frame: Baseline, Week 12 of randomized treatment period
Population: ITT population included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: cm^2
Arm/Group | Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC
Number analyzed (Participants) | 35 | 38
cm^2 | -4.8 [-10.0 to 0.4] | 3.4 [-1.8 to 8.6]
Statistical Analysis 1: Comparison: Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC vs Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC; The mixed model for repeated measures (MMRM) model contained fixed effects for treatment group (categorical variable), visit (ordered categorical variable), and treatment group by visit interaction with additional fixed effects for stratification factors; Test type: Superiority; p = 0.0297, Mixed Models Analysis; Least Square (LS) Mean Difference = -8.2, 95% CI 2-sided [-15.6 to -0.8]

4. Secondary Outcome: Percentage of Participants With New Ulcers by Week 12 in Randomized Treatment Period
Description: New ulcers were defined as ulcer(s) that were not captured at visit 1/screening. In this outcome measure, participants with occurrence of new ulcers during 12 weeks of treatment were considered.
Time Frame: Through Week 12 of randomized treatment period
Population: ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC | Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC
Number analyzed (Participants) | 45 | 43
Percentage of participants | 24.4 [12.9 to 39.5] | 32.6 [19.1 to 48.5]
Statistical Analysis 1: Comparison: Voxelotor (Blinded) + SOC Then Voxelotor (Open Label) + SOC vs Placebo (Blinded) + SOC Then Voxelotor (Open Label) + SOC; Test type: Superiority; p = 0.3456, Cochran-Mantel-Haenszel; Difference in percentage = -8.1, 95% CI 2-sided [-26.9 to 10.7]

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 4 weeks post last dose of study drug: maximum up to approximately 16 weeks for double blinded randomized treatment; maximum up to approximately 89.43 weeks for open label treatment
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as SAE in 1 participant and as non-SAE in another, or a participant may have experienced both the event. Data is reported for study intervention received by participants in the study. Safety-evaluable population included all randomized participants who received at least one dose of study intervention.
Groups:
- Placebo, Blinded: Participants who received placebo matched to voxelotor, orally, once daily for 12 weeks in blinded treatment period.
- Voxelotor, Blinded: Participants who received voxelotor 1500 mg (3 tablets*500 mg) orally, once daily for 12 weeks in blinded treatment period.
- Delayed Voxelotor, Open Label: Participants who received placebo matched to voxelotor, orally, once daily for 12 weeks in blinded treatment period and then who received at least one dose of voxelotor 1500 mg (3 tablets*500 mg) orally, once daily in open label treatment period.
- Voxelotor, Open Label: Participants who received voxelotor 1500 mg (3 tablets*500 mg) orally, once daily for 12 weeks in blinded treatment period and then who received at least one dose of voxelotor 1500 mg (3 tablets*500 mg) orally, once daily in open label treatment period.
Arm/Group | Placebo, Blinded | Voxelotor, Blinded | Delayed Voxelotor, Open Label | Voxelotor, Open Label
All-Cause Mortality (participants affected / at risk) | 0/43 | 1/45 | 4/43 | 6/43
Serious Adverse Events (participants affected / at risk) | 14/43 | 18/45 | 25/43 | 30/43
Other Adverse Events (participants affected / at risk) | 25/43 | 37/45 | 36/43 | 31/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Blinded (N=43) | Voxelotor, Blinded (N=45) | Delayed Voxelotor, Open Label (N=43) | Voxelotor, Open Label (N=43)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 4 (4) | 7 (7) | 5 (5)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 2 (3)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic sequestration (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 4 (4) | 2 (2) | 9 (13) | 10 (12)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 3 (7)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complicated malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis C antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue haemorrhagic fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 9 (9) | 13 (15) | 18 (40) | 23 (40)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Blinded (N=43) | Voxelotor, Blinded (N=45) | Delayed Voxelotor, Open Label (N=43) | Voxelotor, Open Label (N=43)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 4 (5) | 13 (16) | 13 (18) | 10 (17)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (9) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3) | 3 (4) | 4 (5)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Infected skin ulcer (Infections and infestations) | 3 (3) | 0 (0) | 4 (4) | 2 (3)
Malaria (Infections and infestations) | 5 (6) | 5 (6) | 9 (11) | 8 (15)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 8 (8) | 6 (10) | 7 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 5 (7) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 8 (10) | 6 (8) | 6 (9)
Headache (Nervous system disorders) | 3 (3) | 5 (7) | 5 (7) | 3 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 (12) | 8 (11) | 9 (17) | 4 (7)
Venous ulcer pain (Skin and subcutaneous tissue disorders) | 3 (6) | 5 (6) | 4 (5) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-12-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT05561140/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT05561140/SAP_001.pdf